CLINICAL TRIAL: NCT06666985
Title: Intrathecal Morphine for Postoperative Analgesia in Major Laparoscopic Abdominal Surgery (IMPACT-Scope): a Randomised, Sham-controlled, Blinded, Multicentre Clinical Trial
Brief Title: Intrathecal Morphine for Postoperative Analgesia in Major Laparoscopic Abdominal Surgery, a IMPACT-Scope Trial
Acronym: IMPACT-Scope
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT-2023-989
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-12

CONDITIONS: Patients Undergoing Major Laparoscopic Abdominal Surgery
Keywords: laparoscopic surgery; intrathecal morphine; quality of recovery
MeSH Terms: interventions — SLC22A18 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ITM + Usual Care (Experimental)
  Interventions: Drug: ITM + Usual Care
- Sham ITM + Usual Care (Sham Comparator)
  Interventions: Drug: Sham ITM + Usual Care

INTERVENTIONS:
Drug: ITM + Usual Care — The participants allocated to this group will receive ITM (Intrathecal Morphine) in addition to usual care with opioid-based PCA(Patient-Controlled Analgesia). ITM consists of an intrathecal injection of 300 micrograms (0.3mg) of preservative-free morphine.Usual care involves postoperative analgesia with opioid-based PCA without postoperative continuous infusion of opioids. No other drugs other than opioids are allowed in the PCA.
  Arms: ITM + Usual Care
Drug: Sham ITM + Usual Care — The sham ITM mimics the ITM procedure, but the dura is not breached.
  Arms: Sham ITM + Usual Care

SUMMARY:
The goal of this clinical trial is to learn the clinical and cost effectiveness of intrathecal morphine (ITM) in addition to usual care as a postoperative pain relief strategy following major laparoscopic abdominal surgery compared with current usual care. The main questions it aims to answer are:

An enhanced analgesic technique, consisting of ITM in addition to usual care , improves the postoperative quality of recovery at day 1 after surgery by at least 6 points on the 15-item quality of recovery questionnaire (QoR-15) compared to usual care alone, in patients undergoing major laparoscopic abdominal surgery?

Researchers will compare ITM + Usual care to Sham ITM + Usual Care (The sham ITM mimics the ITM procedure, but the dura is not breached) to see if ITM works to postoperative pain relief.

Participants will:

Receive ITM + Usual care or Sham ITM + Usual care on surgery day Have interview with outcome assessors and complete the CRFs on the day of surgery, postoperative day 1, day 2, day 3 and up to postoperative day 30

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or over AND able to give informed consent (with interpreters provided where necessary)
* Elective (i.e., planned) laparoscopic or robotic abdominal surgery within one or more of the following specialties:

  * Colorectal
  * Gynaecology
  * Hepato-biliary (including pancreatic surgery)
  * Upper gastrointestinal
  * Urology/Renal
* Anticipated duration of surgery ≥ 2 hours (from knife-to-skin to end of wound closure)
* Anticipated hospital stay ≥ 24 hours (from the end of surgery)

Exclusion criteria:

* Allergy to study drugs
* Anatomical factors making intrathecal injection impossible
* Anticipated requirement for postoperative invasive ventilation
* American Society of Anesthesiologists (ASA) Score <IV
* Coagulopathies (i.e. INR>1.3 and/or platelet count<100×10^9/L)
* Cognitive impairment leading to inability to complete the study processes and questionnaires
* Drugs affecting coagulation (except aspirin), which have not been suitably and timely paused preoperatively
* Infection near the planned site of intrathecal injection
* Ongoing sepsis
* Patients previously included in the trial and who need to return to theatre for a new abdominal surgery
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | Postoperative day 1
  Quality of recovery is measured using the 15-item Quality of Recovery Questionnaire (QoR-15)

SECONDARY OUTCOMES:
Quality of recovery | Postoperative day 2 , Postoperative day 3 (or at discharge, if earlier)
  Quality of recovery is measured using the 15-item Quality of Recovery Questionnaire (QoR-15)
Quality of life | Postoperative day 1, Postoperative day 2, Postoperative day 3 (or at discharge, if earlier) and Postoperative day 30
  Quality of life is measured using the European Quality of life-5 Dimensions-5 Level (EQ-5D-5L)
Pain scores in the post-anaesthesia recovery unit | Day of surgery
  Pain scores is measured using a numeric rating scale (NRS 0-10)
Worst pain score | Postoperative day 1, Postoperative day 2, and Postoperative day 3 (or at discharge, if earlier)
  Worst pain score is measured using a numeric rating scale (NRS 0-10)
Anaesthesia-related discomfort (nausea and/or vomiting, drowsiness, shivering, pruritus) | Postoperative day 1, Postoperative day 2, Postoperative day 3 (or at discharge, if earlier)
  Anaesthesia-related discomfort is measured using a bespoke questionnaire
Patient satisfaction | Postoperative day 1, Postoperative day 2, Postoperative day 3 (or at discharge, if earlier)
  Patient satisfaction is measured using a bespoke questionnaire
Time in minutes to tracheal extubation from the end of anaesthesia | From end of anesthesia to tracheal extubation on day of surgery or from end of anesthesia to discharge day (for ICU patients) up to 48 hours
Number of pain management visits | Postoperative day 1, Postoperative day 2, Postoperative day 3(or at discharge, if earlier), day of discharge and Postoperative day 30
Postoperative pulmonary complications | Postoperative day 1, Postoperative day 2 and Postoperative day 3 (or at discharge, if earlier)
  Postoperative pulmonary complications is measured according to the Standardized Endpoints for Perioperative Medicine and the Core Outcome Measures in Perioperative and Anaesthetic Care (StEP-COMPAQ) definition
Respiratory depression | Day of surgery, Postoperative day 1, Postoperative day 2, Postoperative day 3 (or at discharge, if earlier)
  Respiratory depression is defined as respiratory rate less than 8 breaths per minute AND need for medical intervention
Total opioid consumption | During operation and up to Postoperative day 30
  Total opioid consumption is transformed into oral morphine equivalent daily dose
Postoperative mobilisation | Postoperative day 1,Postoperative day 2, Postoperative day 3 (or at discharge, if earlier)
  Postoperative mobilisation is ability to transfer from bed to chair, with or without assistance
Doses of antiemetics administered postoperatively (number of administration) | Day of Surgery, Postoperative day 1, Postoperative day 2, Postoperative day 3 (or at discharge, if earlier)
Length of Hospital Stay | 1 Day after surgery
  Length of Hospital Stay (in days) is number of days from starting day of surgery to the day of discharge, calculated as discharge date - surgery date + 1 day
Days at Home and well After Surgery (DAH-30) | Postoperative day 30
Mortality | Postoperative day 30

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China